CLINICAL TRIAL: NCT02304068
Title: The Accuracy of Home Monitoring for Disease Activity During Maintenance Therapy for Neovascular Age-related Macular Degeneration
Brief Title: The Accuracy of Home Monitoring for Acute Macular Degeneration (AMD) Disease Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: OP12/10204; 12/YH/0195 (Other: Research Ethics Committee)
Record Dates: First submitted 2014-11-04; First posted 2014-12-01 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Acute Macular Degeneration
MeSH Terms: interventions — Blood Glucose Self-Monitoring

ARMS (1):
- Intra-vitreal injection (Other)
  Interventions: Other: Home monitoring; Other: Hospital assessment

INTERVENTIONS:
Other: Home monitoring
Other: Hospital assessment

SUMMARY:
Currently the best treatment for "wet" macular degeneration involves regular injections of Ranibizumab (Lucentis). In the initial clinical trials, the drug was injected into the eye every month. Since then a number of studies have found similar benefits when the drug is given with a fixed number of injections initially and then with further injections only when needed. This approach has been adopted in the UK, following recommendation by the National Institute for Clinical Excellence (NICE).

Although this approach reduces the expense and risk of un-necessary treatment, it does require regular hospital assessment of disease activity to determine if a repeat injection is required or can be deferred. The hospital assessment is time-consuming, inconvenient and the large number of assessments can cause delays in hospital follow-up.

Using three different assessment criteria to monitor disease activity at home, the investigators plan to see if home monitoring is as good as hospital assessment. The investigators have already identified that many patients dislike the lengthy hospital assessment visit and would welcome the opportunity to do some of the monitoring of disease activity at home. The investigators have also shown that they understand and can complete each of the home assessment tests. In this pilot project, the investigators aim to get an idea of how reliable home monitoring can be in a small sample of just over 30 patients. The data that the pilot project generates will be used to influence and to help plan a subsequent, larger, national study to be submitted for funding to the National Institute for Health Research.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 60 years with a clinical diagnosis of neovascular age-related macular degeneration (ARMD), receiving treatment with intra-vitreal ranibizumab in accordance with current UK practice
* At least 6 months of prior treatment beyond the loading phase of three fixed injections
* At least 2 injections during the prior 6 months of the maintenance phase of treatment
* Early Treatment for Diabetic Retinopathy Study (ETDRS) chart letter score at 2m of between 30 and 70 letters at the start of the study

Exclusion Criteria:

* Patients with chronic intra-retinal cycts or sub-retinal fluid in the study eye on Optical coherence tomography (OCT) examination despite prior treatment and judged to be stable without the need for further treatment
* Significant hearing impairment, felt likely to interfere with training and the telephone calls prior to the home monitoring
* Lack of informed consent

Ages: 60 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Monitor disease activity at home using near reading chart | 7 months
  The reproducibility of the home monitoring assessment exercise